CLINICAL TRIAL: NCT06612736
Title: Real World Evidence Study: Improving Nutritional Management of Neurologically Impaired Children
Brief Title: Nutritional Management of Neurologically Impaired Children Across China
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Li Hong, Vice President at Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SCMCIRB-K2021078-1
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2021-12

CONDITIONS: Neurological Impairments
Keywords: neurological impairment; enteral nutrition; children; nutritional management
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A retrospective study to (1) investigate clinical characteristics, nutritional status, and nutritional management in neurologically impaired children in China, (2) assess whether enteral nutrition (particularly tube feeding) contributes to improving nutritional outcomes in children with neurological impairments, (3) examine the tolerability of enteral nutrition and whether it can effectively reverse or prevent severe malnutrition.

DETAILED DESCRIPTION:
Electronic health records of children with neurological impairments from 11 medical centers across China between 2015 and 2020 were reviewed. Data were analyzed using SPSS 22.0. Normally distributed data were presented as mean±standard deviation (SD), and non-normally distributed data were presented as median and interquartile range (IQR). Categorical data were presented as frequencies and analyzed using the chi-square test. The Wilcoxon test was used to compare data at different time points. Multivariate logistic regressions were used to analyze the factors influencing gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

(1) age≤18 years, (2) with primary, progressive or non-progressive neurological impairment, (3) received oral nutrition or tube feeding, (4) for tube-fed patients only: at least 1 month of nutritional intervention and at least 1 follow-up visit (i.e. at least at Visit 1)

Exclusion Criteria:

with acquired causes of neurological damage (e.g., traumatic brain injury) or tube-fed patients who received nutritional intervention for less than a month and without follow-up

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with neurological impairments across China
Sampling Method: Non-Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Weight for age z-score | From diagnosis to 24 months of follow-up
  It indicates body weight of a children for their age and sex relative to the reference population. It is an important indicator of acute nutritional status in young children aged less than two years old.
Height for age z-score | From diagnosis to 24 months of follow-up
  It indicates height of a children for their age and sex relative to the reference population. It is an important indicator of chronic nutritional status in children.
BMI for age z-score | From diagnosis to 24 months of follow-up
  It indicates body mass index of a children for their age and sex relative to the reference population. It is an important indicator of acute nutritional status in children aged greater than two years old.

CONTACTS AND LOCATIONS:
Overall Officials: Li Hong, MD, PhD, Principal Investigator — Shanghai Children's Medical Center Affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- Shanghai Children's Medical Center Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided